CLINICAL TRIAL: NCT00539643
Title: A Randomized Single Blind Controlled Trial of Beads vs. Doxorubicin Eluting Beads for Arterial Embolization of Hepatocellular Carcinoma (HCC)
Brief Title: Trial of Beads Versus Doxorubicin Eluting Beads for Arterial Embolization of Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-099
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Hepatoma
Keywords: Liver Cancer; Hepatoma; 07-099
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Bead Arm (Active Comparator): Hepatic arterial embolization with Bead Block microspheres, beginning with 100 - 300 micron beads, and using larger particles if necessary until stasis is evident.
  Interventions: Device: Bead Block microspheres
- Bead + Dox Arm (Active Comparator): Hepatic arterial embolization with 100-300 micron drug eluting microspheres (LC Bead) loaded with 150 mg Doxorubicin, followed by embolization with Bead Block microspheres (100-300 micron and larger size beads as necessary) until stasis is evident.
  Interventions: Other: Bead + Dox Arm

INTERVENTIONS:
Device: Bead Block microspheres — Bead Block (Beads) microsphere, 100-300 micron with additional larger size beads as necessary to achieve stasis
  Arms: Bead Arm
Other: Bead + Dox Arm — Bead + Dox Arm: Hepatic arterial embolization with 100-300 micron drug eluting microspheres (LC Bead) loaded with 150 mg Doxorubicin, followed by embolization with Bead Block microspheres (100-300 micron and larger size beads as necessary) until stasis is evident.
  Arms: Bead + Dox Arm

SUMMARY:
The purpose of this study is to evaluate the effect of blocking the blood vessels to the tumor in your liver with small beads alone (Bead Block) versus blocking them with the same bead that contains and releases doxorubicin (a chemotherapy agent). The reason for the study is to see if adding doxorubicin kills more tumor than would be killed by just blocking the blood supplying the tumor. The chemotherapy, doxorubicin, has been used for many years to treat patients with cancer. This procedure to block the blood vessels is called embolization. Embolization is a common treatment for patients with liver cancer who cannot have surgery. The investigators are comparing the standard treatment (using the small beads alone) with another that should be at least as good, but possibly better (with the addition of the drug, doxorubicin). There is no guarantee that the new treatment is better and it is possible that there might be more side effects (related to the doxorubicin) than what is seen with the standard treatment.

DETAILED DESCRIPTION:
Biocompatibles LC Bead (also known as DC Bead in Asia & Europe) microspheres are preformed soft, deformable microspheres that may be loaded with doxorubicin and used to occlude blood flow to a cancerous tumour. LC Bead microspheres consist of a macromere derived from PVA. The fully polymerized microsphere is approximately 90% water and is compressible to approximately 30% by diameter. The microspheres can be delivered through conventional catheters (4-5Fr) or micro-catheters in the 2-3Fr range. These microspheres, like all agents used for arterial embolization, are mixed with radiographic contrast prior to administration in order to allow for fluoroscopic control of the embolization procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a confirmed diagnosis of HCC according to EASL criteria for diagnosis; who is not a surgical resection candidate, or refuses surgery
* Patient must be 18 years of age or older
* Patient must be Okuda stage I or II
* Patient must have an ECOG performance status of 0 or 1
* No prior chemotherapy or biotherapy within 4 weeks of scheduled embolization, with all toxicities, if any, resolved to grade < than or = to 1
* Patient must have the following laboratory values confirmed within 14 days of registration:
* Creatinine ≤ than or = to 2.0 the institution ULN
* Platelets ≥ than or = to 50,000/mm3
* INR ≤ than or = to 2.0 for patients who are not on Coumadin
* aPTT < or = to twice control
* Bilirubin < 3 mg/dl
* WBC > 3000 cells/mm3
* ANC > 1500 cells/mm3
* Negative serum pregnancy test (Female of childbearing potential only)

Exclusion Criteria:

* Patient has another primary tumor, with the exception of conventional basal cell CA, superficial bladder cancer, melanoma in situ, or treated prostate cancer currently without biochemical or radiographic evidence of active disease
* Women who are pregnant or lactating
* Patient previously treated with doxorubicin
* Contraindication to angiography/embolization including: patients who cannot receive contrast 1.Severe allergic reaction to contrast despite pre-medication, 2. poor renal function; 3.Lack of arterial access (eg femoral artery occlusion); 4. other, based on judgment of the investigator
* Patient has already undergone hepatic arterial embolization for the hepatocellular cancer for which they are currently being evaluated
* Patient has received prior radiotherapy for the hepatocellular cancer for which they are currently being evaluated
* Patient has had previous local-regional treatment of the current target tumor volume
* Patient who cannot have CT scan
* Patient at very high risk for post-embolization hepatic failure: 1. Child's C cirrhosis, 2. > 75% liver replaced by tumor
* Cardiac exclusion for: 1. Myocardial infarction within 90 days of study, 2. uncontrolled arrhythmia, 3. LVEF < 50% for patients randomized to receive LC Bead
* Patients with tumors exhibiting characteristics considered contra-indications to particle embolization, including: 1. collateral vessel pathways potentially endangering normal territories during embolization, 2. arteries supplying tumor not large enough to accept LC Bead or Bead Block, 3. Presence of arterial to systemic venous shunts, 4. Presence of arterial to pulmonary vascular shunts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen T Brown, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Brown KT, Do RK, Gonen M, Covey AM, Getrajdman GI, Sofocleous CT, Jarnagin WR, D'Angelica MI, Allen PJ, Erinjeri JP, Brody LA, O'Neill GP, Johnson KN, Garcia AR, Beattie C, Zhao B, Solomon SB, Schwartz LH, DeMatteo R, Abou-Alfa GK. Randomized Trial of Hepatic Artery Embolization for Hepatocellular Carcinoma Using Doxorubicin-Eluting Microspheres Compared With Embolization With Microspheres Alone. J Clin Oncol. 2016 Jun 10;34(17):2046-53. doi: 10.1200/JCO.2015.64.0821. Epub 2016 Feb 1. PMID 26834067
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bead Arm | Bead + Dox Arm
Started | 51 | 50
Completed | 45 | 47
Not Completed | 6 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Death | 2 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bead Arm | Bead + Dox Arm | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Full Range); unit: years] | 68 [41 to 87] | 66 [29 to 86] | 67 [29 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 37 | 41 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 51 | 50 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 41 | 38 | 79
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment by RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bead Arm | Bead + Dox Arm
Number analyzed (Participants) | 51 | 50
Participants
  Participants With Response | 3 | 3
  Participants Without Response | 48 | 47

2. Secondary Outcome: Number of Participants Evaluated for Toxicity
Description: Toxicity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) 3.0.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bead Arm | Bead + Dox Arm
Number analyzed (Participants) | 51 | 50
Participants | 51 | 50

3. Secondary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year
Measure: Median (Standard Deviation); unit: months
Arm/Group | Bead Arm | Bead + Dox Arm
Number analyzed (Participants) | 51 | 50
months | 6.2 (.11) | 2.8 (.11)

4. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bead Arm | Bead + Dox Arm
Number analyzed (Participants) | 51 | 50
Participants
  Alive | 3 | 3
  Dead | 48 | 47

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bead Arm | Bead + Dox Arm
All-Cause Mortality (participants affected / at risk) | 48/51 | 47/50
Serious Adverse Events (participants affected / at risk) | 48/51 | 47/50
Other Adverse Events (participants affected / at risk) | 33/51 | 28/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bead Arm (N=51) | Bead + Dox Arm (N=50)
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Liver abscess (Hepatobiliary disorders) | 1 | 0
Liver failure (transient) (Hepatobiliary disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Puncture Site (Injury, poisoning and procedural complications) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Pulmonary embolus (Vascular disorders) | 1 | 4
Death not assoc w CTCAE term- Death (General disorders) | 3 | 4
Death not assoc w CTCAE term- Sudden death (General disorders) | 1 | 0
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 4 | 5
Death due to disease progression (General disorders) | 40 | 38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bead Arm (N=51) | Bead + Dox Arm (N=50)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Alkaline Phosphatase (Investigations) | 9 | 9
Allerg react/hypersens (incl drug fever) (Immune system disorders) | 1 | 0
ALT, SGPT (Investigations) | 14 | 11
Amylase (Investigations) | 1 | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 3 | 2
AST, SGOT (Investigations) | 7 | 6
Atrial fibrillation (Cardiac disorders) | 2 | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 4 | 11
Blood/Bone Marrow, other (Blood and lymphatic system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 1
Creatinine (Investigations) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 | 3
Fever (in the absence of neutropenia) (General disorders) | 4 | 3
Gastritis (incl bile reflux gastritis) (Gastrointestinal disorders) | 0 | 1
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 5 | 6
Hemoglobin (Blood and lymphatic system disorders) | 2 | 1
Hemorrhage, Lower GI NOS (Gastrointestinal disorders) | 1 | 0
Hemorrhage, Rectum (Gastrointestinal disorders) | 1 | 0
Hemorrhage, Varices (esophageal) (Gastrointestinal disorders) | 1 | 1
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 1 | 0
Hepatobiliary/Pancrease, other (Hepatobiliary disorders) | 1 | 0
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ileus, GI (func obstruction of bowel) (Gastrointestinal disorders) | 2 | 1
Inf norm ANC/gr1/2 neut- Pneumonia(lung) (Investigations) | 1 | 0
Inf unknown ANC-Cellulitis(skin) (Infections and infestations) | 0 | 1
Infection w/ Gr 3/4 neut, Urinary tract NOS (Infections and infestations) | 1 | 0
INR (Investigations) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Leak, GI- Biliary tree (Gastrointestinal disorders) | 1 | 0
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 | 2
Lipase (Investigations) | 0 | 1
Liver dysfunction/failure (Hepatobiliary disorders) | 2 | 6
Lymphopenia (Investigations) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT00539643/Prot_SAP_000.pdf